CLINICAL TRIAL: NCT06429813
Title: A Feasibility Study to Examine the Impact of Remotely Monitored Exercise Interventions on Cardiorespiratory/muscular Fitness and Fatigue in Patients with Metastatic Castrate-sensitive Prostate Cancer (mCSPC) Undergoing Treatment with Androgen-deprivation Therapy (ADT) Intensification
Brief Title: Remotely Monitored Exercise Interventions in Patients with MCSPC Undergoing ADT (Prostate 006)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Viscuse (Other)
Responsible Party: Sponsor-Investigator, Paul Viscuse, Assistant Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR230542
Record Dates: First submitted 2024-05-14; First posted 2024-05-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-08

CONDITIONS: Castrate Sensitive Prostate Cancer; Metastatic Prostate Cancer
Keywords: prostate; metastatic prostate cancer; metastatic castrate-sensitive prostate cancer; prostate cancer; exercise; ADT; ARSI
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): HIIT Cycling Intervention
  Interventions: Behavioral: Home-Based Exercise Intervention - HIIT Cycling
- Arm B (Experimental): Walking Intervention
  Interventions: Behavioral: Home-Based Exercise Intervention - Walking

INTERVENTIONS:
Behavioral: Home-Based Exercise Intervention - Walking — 30 minutes of walking or light jogging a day at a moderate intensity for 30 minutes a day, 5 days a week for 12 weeks
  Arms: Arm B
Behavioral: Home-Based Exercise Intervention - HIIT Cycling — Four, 4 minute high intensity intervals of exercise, separated by 3 minutes of lower intensity exercise + a 10 minute warm up and 5 minute cool down for 40 minutes a day, 3 days a week for 12 weeks
  Arms: Arm A

SUMMARY:
This study consists of two home-based exercise programs: a stationary exercise bicycle intervention (Arm A), and a walking intervention (Arm B). The study will enroll 24 patients who are starting ADT (Androgen Deprivation Therapy)/ARSI (Androgen-Receptor Signaling Inhibitors) therapy for newly diagnosed metastatic castrate-sensitive prostate cancer (mCSPC). All participants will be asked to complete 1-2 training sessions at UVA prior to starting the exercise. All participants will be asked to complete aerobic and strength testing before and after the exercise program. Participants will be asked to answer questionnaires throughout the program. The at-home exercise will last for 12 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to find out how many patients who are being treated for mCSPC complete one of two home-based exercise programs. The researchers want to find out how much exercise participants complete and how satisfied they are with the program. Another purpose of this study is to learn if doing the exercise changes fitness levels and/or muscle strength, and what relationship those changes might have on feeling tired during cancer treatment.

Participants will be randomly assigned (like the flip of a coin) to one of two home-based exercise programs:

* Arm A: A high intensity interval (HIIT) stationary bike program
* Arm B: A walking program

Participants in the cycling group (Arm A) will receive a stationary exercise bike for home exercise. All participants in the study (Arms A and B) will receive an activity monitor (watch) and a heart rate-monitoring chest strap that sends information back to the study team.

Participants will receive 1-2 exercise training sessions, held in a UVA research lab, to allow them to experience the level of the exercise they will be asked to complete. Each participant will make a personal plan with the study team to gradually workup to the exercise goal assigned to each group. The research team will answer any questions and help set up the activity monitors. After these session(s), the remaining 12 weeks of exercise will occur at home.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male, aged ≥18 years old
4. Diagnosis of mCSPC (defined as either biopsy-proven metastatic prostate cancer or elevated PSA (Prostate Specific Antigen) in the setting of imaging findings typical of prostate cancer spread; patients can either have de novo metastatic disease or recurrent metastatic disease after prior definitive therapy to the primary tumor with either surgery or radiation)
5. Planned treatment with ADT (LHRH [Luteinizing hormone-releasing hormone] agonist such as leuprolide or LHRH antagonist such as degarelix), or recent administration, ≤14 days prior to enrollment.
6. Planned intensification with ARSI (abiraterone/prednisone, enzalutamide, apalutamide, or darolutamide).
7. Oncologist clearance for exercise training after taking into account functional status and co-morbid conditions that may limit ability to participate.
8. Ability to take oral medication and willing to adhere to the study intervention regimen
9. Ability to read, speak, and understand English.

Exclusion Criteria:

1. Castrate-resistant prostate cancer (defined as prostate cancer previously treated with a backbone of ADT hormonal therapy with either progression of disease on imaging PSA progression with PSA increase of > 25% and 2 ng/mL above nadir, confirmed at 2 time points at least 3 weeks apart, in the setting of testosterone level < 50)
2. Patients with prostate cancer with biochemical recurrence (e.g., received prior definitive therapy with subsequent PSA [Prostate-Specific Antigen] rise) but radiographic imaging is negative for metastatic disease
3. Metastatic bone lesion(s) in the proximal femur, bone lesion causing impending fracture, or other metastatic site deemed unsafe for walking by treating physician
4. Medical/orthopedic comorbidities that preclude stationary cycling or walking
5. Significant cardiac/renal/hepatic/hematological/pulmonary disease precluding exercise training
6. Unstable angina or myocardial infarction within 4-weeks prior to treatment
7. Complex ventricular arrhythmias or New York Heart Association class IV symptoms
8. Symptomatic severe aortic stenosis
9. Acute pulmonary embolus
10. Acute myocarditis
11. Untreated high-risk proliferative retinopathy
12. Recent retinal hemorrhage
13. Uncontrolled hypertension (systolic blood pressure > 180 mm Hg or diastolic blood pressure > 120 mm Hg)
14. Severe baseline electrolyte abnormalities (e.g. potassium) that may predispose patient to arrhythmias in the opinion of the treating investigator
15. Uncontrolled metabolic disease (diabetes with fasting blood sugar >300 mg/dl, thyrotoxicosis, myxedema)
16. Symptomatic peripheral vascular disease
17. Prior treatment with taxane- or platinum- based chemotherapy
18. Prior treatment with PARP [Poly (ADP-ribose) polymerase] inhibitors
19. Prior treatment with radium-223 or lutetium-177

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete the post-intervention follow-up assessment | 14 weeks from the start of the intervention
  Percentage of participants who complete the post-intervention follow-up assessment

SECONDARY OUTCOMES:
Treatment engagement with intervention | From the beginning of the intervention to the Post-intervention visit (about 12 weeks)
  Frequency, intensity and duration of exercise as measured by the activity monitors.
Acceptability of exercise | From the beginning of the intervention to the Post-intervention visit (about 12 weeks)
  The Physical Activity Enjoyment Scale (PACES) is an 18 question, 7 point scale that includes questions regarding enjoyment of physical activity in the study.
Patient-reported outcomes on exercise | From the beginning of the intervention to the Post-intervention visit (about 12 weeks)
  Exit interviews include open and closed ended questions about the participant's experience in the study.
Rate of recruitment per month | Each month for 12 months (estimated duration of accrual of participants)
  Number of individuals screened and randomized
Physical fitness (Cardiorespiratory) | Measured at the baseline visit before the start of the intervention and post-intervention visit (about 16 weeks later)
  As measured by VO2 peak
Muscular strength (quadriceps) | Measured at the baseline visit before the start of the intervention and post-intervention visit (about 16 weeks later
  Isometric and isokinetic torque in multiple positions (e.g. 60-120 degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Viscuse, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No